CLINICAL TRIAL: NCT01702662
Title: The Assessment of the Photopill Capsule Treatment for Safety and Feasibility in Healthy Volunteers, a Phase 1 Trial
Brief Title: Photopill Treatment in Healthy Volunteers
Acronym: Photopill
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Hanke Brandse, MD, Phd student, executive investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: METC2012_150, ABR: 40642
Record Dates: First submitted 2012-10-03; First posted 2012-10-08 (Estimated); Last update posted 2012-12-11 (Estimated); Status verified 2012-12

CONDITIONS: Ulcerated Mucosa of Colon

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Photopill treatment (Experimental): Photopill treatment, 2 minutes per cm rectal mucosa (3cm) 10 times
  Interventions: Device: Photopill treatment

INTERVENTIONS:
Device: Photopill treatment — 2 courses of 5 Photopill treatments within 14 days. In each treatment, 3cm of rectal tissue will be exposed, 2 minutes per cm, to low level light therapy.

SUMMARY:
Photo-bio-stimulation by Low Level Light therapy(LLLT) has demonstrated its clinical use in chemotherapy/radiotherapy oral mucositis.

Unpublished study (Melzer, Ben-Yehuda et al. UEGW 2012) with the Photopill (LLLT) capsule treatment in mice showed a significant beneficial effect on the endoscopic severity of DSS-induced colitis in mice.

Therefore a phase 1 trial is designed to assess the safety and feasibility of the Photopill treatment in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are generally healthy.
* Signed informed consent.

Exclusion Criteria:

* Subjects with any known GI related symptoms complaints or GI diseases.
* Subjects with cancer or other life threatening diseases or conditions.
* Subjects with cardiovascular or pulmonary diseases.
* Pregnant women.
* Subjects who underwent any colon surgery.
* Morbid Obesity (BMI > 40).
* Drug abuse or alcoholism.
* Bed-ridden patient.
* Any rectal therapy.
* Participation in current clinical study or clinical study within 30 days prior to the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2012-08; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (Mucosal Aspect at 2nd sigmoidoscopy after 7-14 days) as a Measure of Safety and Tolerability | During Study period: day 0-14

CONTACTS AND LOCATIONS:
Overall Officials: Geert D'Haens, Prof.dr, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Academic Medical Center Amsterdam, department of Gastroenterology, Amsterdam, North Holland, Netherlands